CLINICAL TRIAL: NCT00796159
Title: A Post Marketing Surveillance, Multicenter, Open-Label, Dose-Titrating, 4-Week Study Evaluating The Efficacy, Tolerability And Safety Of Olmesartan Medoxomil 20mg In Combination With 12.5mg Hydrochlorothiazide In Subjects With Stage 1 To Stage 2 Hypertension
Brief Title: Post-Marketing Surveillance Of Olmesartan Medoxomil In Combination With Hydrochlorothiazide
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A0021004
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: Efficacy; Tolerability; Safety; Essential Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Olmesartan medoxomil + HCTZ
  Interventions: Drug: Olmesartan medoxomil

INTERVENTIONS:
Drug: Olmesartan medoxomil — olmesartan medoxomil 20 mg and HCTZ 12.5 mg

SUMMARY:
This is a Post-Marketing Surveillance study evaluating the Efficacy, Tolerability and Safety of Olmesartan medoxomil 20 mg in combination with 12.5 MG of hydrochlorothiazide in subjects with mild to moderate essential hypertension

DETAILED DESCRIPTION:
Non Probability Sampling

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients 18 to 65 y/old
* Patient previously taking low-dose medoxomil or any other ARB alone with uncontrolled BP
* Patient with uncontrolled mild to moderate hypertension (SBP>= 140 and <=179 mmHg OR DBP of >=90 and <=109 mmHg)

Exclusion Criteria:

* Pregnant of Lactating women
* History of secondary hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino patients with Uncontrolled Mild to Moderate Essential Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1723 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse Events) | 4 weeks

SECONDARY OUTCOMES:
Blood Pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0021004&StudyName=Post-Marketing%20Surveillance%20Of%20Olmesartan%20Medoxomil%20In%20Combination%20With%20Hydrochlorothiazide%20